CLINICAL TRIAL: NCT06982898
Title: Restorative Comparison of Facebow and Simplified Techniques for Digital Jaw Relation Records in Treatment of Occlusal Rehabilitation
Brief Title: Digitalization of Maxillo-mandibular Relation for Arches With Occlusal Support Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kıvanç Akça (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Kıvanç Akça, Professor, Department of Prosthodontics, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA-24002
Record Dates: First submitted 2025-04-21; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Prosthetic Treatment; Occlusal Analysis; Digitalism
Keywords: jaw relation; digital dentistry

STUDY DESIGN:
Intervention Model Description: All participants will receive two different prosthetic interventions based on different jaw relation record techniques. The outcomes will be compared within the same individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determination of Intermaxillary Relationship in Patients with Posterior Support Loss (Experimental): For each participant, an intraoral scan was initially obtained using the bimanual manipulation method to determine the centric relation. Subsequently, the neuromuscular deprogramming method was applied, and recordings were obtained using a jaw movement tracking and analysis device.
  During occlusal adjustment of the restorations fabricated based on both recording methods, the following parameters were evaluated: occlusal surface adaptation, adjustment time, and number of articulating paper applications.
  Interventions: Procedure: Fixed prosthesis with bimanual CR and intraoral scan

INTERVENTIONS:
Procedure: Fixed prosthesis with bimanual CR and intraoral scan — Tooth-supported fixed prostheses were fabricated using centric relation records obtained by two different methods:
  1. Bimanual manipulation technique, with jaw relation records captured using an intraoral scanner.
  2. Neuromuscular deprogramming technique, with jaw relation records obtained using a jaw movement tracking and analysis device.
  Other Names: Fixed prosthesis with neuromuscular CR and jaw tracking

SUMMARY:
Accurate recording of the intermaxillary relationship is crucial for achieving successful restorative outcomes.

In cases of occlusal support loss, determining and recording the intermaxillary relationship becomes more complex.

This study aims to compare the occlusal compatibility of restorations fabricated using either an intraoral scanner or a jaw motion tracking and analysis device for recording the intermaxillary relationship in patients with occlusal support loss.

DETAILED DESCRIPTION:
This study is designed to fabricate bilateral fixed prosthetic restorations in the maxillary posterior region and to evaluate the clinical success, efficiency, and patient satisfaction associated with different intermaxillary relationship recording methods.

The study will compare the clinical outcomes of restorations produced using two techniques:

Group I: Centric relation (CR) determined by bimanual manipulation and recorded with an intraoral scanner.

Group II: Centric relation (CR) determined by neuromuscular deprogramming and recorded with a jaw movement/tracking analysis device.

All tooth preparations will follow standard preparation principles, ensuring minimum material thickness. Preparations will be completed by the investigator (ESK). After preparation, intraoral scans of the upper and lower jaws will be obtained using an intraoral scanner.

Centric relation will be recorded first with bimanual manipulation stabilized with wax, then digitized via intraoral scanning. In a subsequent session, centric relation will be recorded using a neuromuscular deprogrammer and jaw movement tracking analysis.

Both recordings will be sent to a dental laboratory for the fabrication of restorations. A randomization protocol will be applied to vary the adjustment order of the restorations fabricated by each method.

During clinical evaluation:

Distal and mesial proximal contacts will be checked and adjusted as needed.

Internal fit will be evaluated and corrected if necessary.

Occlusal adjustment will be performed using 100 µm and 40 µm articulation papers (Arti-Check micro-thin, Bausch, Cologne, Germany).

After occlusal adjustment:

The adjusted surfaces will be colored, photographed, and measured using ImageJ software to determine the adjusted surface area (in mm²).

Adjustment time and number of articulation paper applications will also be recorded.

These clinical parameters (adjusted area, adjustment time, and number of papers used) will be scored to assess the clinical success of the restorations.

Additionally, patient-reported outcomes will be collected:

Occlusal comfort and technique preference will be evaluated via a Visual Analog Scale (VAS, 0 = complete dissatisfaction, 10 = complete satisfaction) and a method preference survey.

This evaluation aims to determine which technique offers better patient comfort and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation after reading and understanding the informed consent form.
* Age between 18 and 65 years with completed growth and development.
* Healthy dental and periodontal condition.
* Presence of bilateral edentulism in the maxillary posterior region leading to occlusal support loss, requiring fixed prosthetic treatment.
* Fixed dentition present in the mandible.

Exclusion Criteria:

* Refusal to voluntarily participate after reading the informed consent form.
* General health condition unsuitable for prosthetic treatment.
* Use of removable prostheses in the mandibular arch.
* Presence of temporomandibular joint dysfunction, orofacial pain, or acute oral disease.
* Presence of a pacemaker or implantable defibrillator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Adjustment Time for Restoration | 1 year
  The time required to adjust the restoration will be recorded in minutes and scored on a 0-4 scale as follows: 0 (≤1 min), 1 (1-5 min), 2 (5-10 min), 3 (10-15 min), 4 (≥15 min).
Adjusted Surface Area of the Restoration | 1 year
  The surface area requiring adjustment will be measured in square millimeters (mm²) using ImageJ software and scored from 0 to 4: 0 (≤1 mm²), 1 (1-6 mm²), 2 (6-10 mm²), 3 (10-15 mm²), 4 (≥15 mm²).
Number of Articulation Paper Uses | 1 year
  The number of articulation paper uses will be counted and scored from 0 to 4 as follows: 0 (2-4 uses), 1 (5-7), 2 (8-10), 3 (10-13), 4 (≥14 uses).
Composite Clinical Success Score of the Restoration | 1 year
  The clinical success of each restoration will be evaluated using a composite score derived from three parameters:
  Adjustment Time, Adjusted Surface Area,Number of Articulation Paper Uses.
  Each parameter is scored from 0 to 4, yielding a total score between 0 and 12. Based on the total score, restorations will be categorized as follows:
  Excellent (Score 0-1): Restoration has a clinically optimal fit. Occlusal contacts are properly and evenly distributed.
  Successful (Score 2-4): Restoration shows good clinical fit with minor occlusal adjustments.
  Moderate (Score 5-7): Restoration is clinically acceptable with occlusal adjustments.
  Weak (Score 8-10): Restoration has issues in clinical fit and required major occlusal adjustments.
  Unsuccessful (Score 11-12): Clinical fit is unacceptable. Adjustments caused morphological distortion or resulted in occlusal gaps. Restoration must be replaced.
  This composite score will serve as the primary measure of overall clinical success.

SECONDARY OUTCOMES:
Occlusal Comfort Evaluated Using Visual Analog Scale | 1 year
  Secondary outcome will assess patient-reported occlusal comfort following the clinical application of the restoration. Occlusal comfort will be measured using a 10-point Visual Analog Scale (VAS), where 0 indicates no comfort and 10 indicates maximum comfort. Patients will rate their experience immediately after the restoration trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the study focuses on clinical and patient reported outcomes that are not structured for external distribution.

REFERENCES:
- [Background] Jasz B, Ambrus S, Garay T, Schmidt P, Hermann P, Kormendi S, Jasz M. Different methods of determining centric relation - comparison with a digital mandibular motion analyser. BMC Oral Health. 2024 Mar 18;24(1):345. doi: 10.1186/s12903-024-04131-x. PMID 38500122
- [Background] Manfredini D, Ercoli C, Poggio CE, Carboncini F, Ferrari M. Centric relation-A biological perspective of a technical concept. J Oral Rehabil. 2023 Nov;50(11):1355-1361. doi: 10.1111/joor.13553. Epub 2023 Jul 11. PMID 37394665
- [Background] Revilla-Leon M, Fernandez-Estevan L, Barmak AB, Kois JC, Perez-Barquero JA. Accuracy of the maxillomandibular relationship at centric relation position recorded by using 3 different intraoral scanners with or without an optical jaw tracking system: An in vivo pilot study. J Dent. 2023 May;132:104478. doi: 10.1016/j.jdent.2023.104478. Epub 2023 Mar 6. PMID 36889536
- [Background] Revilla-Leon M, Zeitler JM, Kois DE, Kois JC. Utilizing an additively manufactured Kois deprogrammer to record centric relation: A simplified workflow and delivery technique. J Prosthet Dent. 2024 Jul;132(1):20-25. doi: 10.1016/j.prosdent.2022.04.034. Epub 2022 Aug 5. PMID 35934572
- [Background] Radu M, Radu D, Abboud M. Digital recording of a conventionally determined centric relation: A technique using an intraoral scanner. J Prosthet Dent. 2020 Feb;123(2):228-231. doi: 10.1016/j.prosdent.2018.12.004. Epub 2019 May 16. PMID 31104810
- [Background] Abdulateef S, Edher F, Hannam AG, Tobias DL, Wyatt CCL. Clinical accuracy and reproducibility of virtual interocclusal records. J Prosthet Dent. 2020 Dec;124(6):667-673. doi: 10.1016/j.prosdent.2019.11.014. Epub 2020 Feb 1. PMID 32014284
- [Background] Kordass B, Gartner C, Sohnel A, Bisler A, Voss G, Bockholt U, Seipel S. The virtual articulator in dentistry: concept and development. Dent Clin North Am. 2002 Jul;46(3):493-506, vi. doi: 10.1016/s0011-8532(02)00006-x. PMID 12222093
- [Background] Kattadiyil MT, Alzaid AA, Campbell SD. What Materials and Reproducible Techniques May Be Used in Recording Centric Relation? Best Evidence Consensus Statement. J Prosthodont. 2021 Apr;30(S1):34-42. doi: 10.1111/jopr.13321. PMID 33783085